CLINICAL TRIAL: NCT01738633
Title: Quality of Life After Esophagectomy for Cancer - Step 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Surgical Unit closed and moved.
Sponsor: University of Padova (Other)
Collaborators: Fondazione Guido Berlucchi (Other); Veneto Institute of Oncology I.O.V.-I.R.C.C.S. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QOLEC1 - step 2
Record Dates: First submitted 2012-10-20; First posted 2012-11-30 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Esophageal Cancer; Quality of Life
Keywords: Esophageal Cancer; Quality of Life
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- nutritional + respirology counseling (Experimental): patients will receive both nutritional and respirology counseling
  Interventions: Behavioral: nutritional counseling; Behavioral: respirology counseling
- nutritional counseling (Experimental): patients will receive nutritional counseling alone
  Interventions: Behavioral: nutritional counseling
- respirology counseling (Experimental): patients will receive respirology counseling alone
  Interventions: Behavioral: respirology counseling
- standard care (No Intervention): patients will receive standard care

INTERVENTIONS:
Behavioral: nutritional counseling
  Arms: nutritional + respirology counseling; nutritional counseling
Behavioral: respirology counseling
  Arms: nutritional + respirology counseling; respirology counseling

SUMMARY:
Background: A recent systematic review showed that patients undergoing esophagectomy for cancer had scores of physical function, vitality and performance of health in general significantly lower than those obtained from the reference population. The analysis of the quality of life at six months follow-up showed that the total score and physical function were better before surgery and symptoms-based scales indicated that the fatigue, dyspnoea and diarrhea were worse six months after esophagectomy. The objective of this study is therefore to assess the impact of esophageal resections for cancer on the quality of life of patients and to improve it through simple interventions of post operative care.

The study is divided into two steps.

This is step 2.

At hospital discharge, patients will be randomized into 4 groups receiving respectively: nutritional and respirology counseling; nutritional counseling alone; respirology counseling alone; standard care. All the patients fill in the questionnaires QLQ C30, OES18, INPAT32 at 1 and 3 months after the surgical operation. Primary end-points are the items DY (dyspnoea), AP (appetite loss) and QL2 of QLQ C30. Secondary end point is the item EA (eating) of OES18.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years old
* scheduled for esophagectomy for cancer

Exclusion Criteria:

* age below 18 years old
* incapability to autonomously fill in questionnaires
* primary language not italian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
items DY (dyspnoea), AP (appetite loss) and QL2 of the QLQ C30 | 1 month after surgical operation

SECONDARY OUTCOMES:
item EA (eating) of OES18 | 1 month after surgical operation
items DY (dyspnoea), AP (appetite loss) and QL2 of the QLQ C30 | 3 months after surgical operation
item EA (eating) of OES18 | 3 months after surgical operation

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto (IOV-IRCCS), Padua, Italy